CLINICAL TRIAL: NCT04916535
Title: Observational Cohort Prospective Multicenter Study on Mitral Annular Disjunction (MAD) - MAD multiceNter Study (MAD-NesS)
Brief Title: Prospective Multicenter Study on Mitral Annular Disjunction
Acronym: MAD-NesS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital of Ferrara (Other)
Responsible Party: Principal Investigator, Gianluca Campo, Full Professor Cardiologist, University Hospital of Ferrara
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 367/2021/Oss/AOUFe
Record Dates: First submitted 2021-06-03; First posted 2021-06-07 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Mitral Valve Disease
Keywords: mitral annular disjunction

STUDY DESIGN:
Intervention Model Description: Observational cohort prospective multicenter study on patients with MAD
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- diagnostic flow (Experimental): all patients with MAD as assessed during routine transthoracic echocardiography will undergo to the following further exams: i) 12-lead electrocardiogram (ECG), ii) 24-hour ECG monitoring, iii) cardiac magnetic resonance imaging (CMR), iv) cardiological visit
  Interventions: Other: diagnostic flow

INTERVENTIONS:
Other: diagnostic flow — exams to estimate the risk of adverse events in patients with MAD

SUMMARY:
Observational cohort prospective multicenter study on patients with mitral annular disjunction (MAD). MAD is defined as a separation (≥1 mm) between the atrial wall-mitral valvular junction and the left ventricular free wall during end-systole

DETAILED DESCRIPTION:
Mitral annular disjunction (MAD) is a structural abnormality of the mitral annulus, defined as a separation (≥1 mm) between the atrial wall-mitral valvular junction and the left ventricular free wall during end-systole. This abnormality is significantly associated with the presence of mitral valve prolapse (MVP), but it can also be observed in normal hearts. MAD-related hypermobility of the mitral apparatus and the consequent posterior systolic curling determine a mechanical stress of the infero-basal wall and papillary muscle. This phenomenon leads to myocardial hypertrophy and fibrosis, creating an arrhythmogenic substrate and a source of electrical instability. For this reason, the analysis of left ventricle by cardiac magnetic resonance plays a pivotal role in the identification of predictors of fatal arrhythmic events, such as sudden cardiac death (SCD). Taking into account that MAD could be present without MVP, some studies analyzed the association between MAD and arrhythmic events. They showed that MAD itself is a risk marker of electrical instability supporting the existence of an emerging clinical entity: the MAD arrhythmic syndrome. An in deep analysis of MAD patients and their characteristics in terms of EKG, types of arrhythmia, echocardiographic parameters and cardiac magnetic resonance (CMR) data and long-term events is lacking.

The present study is ideated and conducted to fill this gap and collect information regarding management and outcome of patients with MAD

ELIGIBILITY:
Inclusion criteria:

* Subject aged ≥18 years and <65 years
* Evidence of MAD during routine echocardiography clinically indicated by treating physician for any reason
* Written informed consent

Exclusion criteria:

• Patient's refusal

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 249 (Actual)
Dates: Start 2021-06-03 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2030-07-01 (Estimated)

PRIMARY OUTCOMES:
Pathological findings associated with MAD | 3 months
  Percentage of subjects with MAD whom deeper analysis with cardiological visit, electrocardiogram (ECG), 24-hour ECG Holter monitoring and cardiac magnetic resonance (CMR) identifies pathological findings. Pathological findings are defined as follows: -T wave inversion in inferolateral leads at ECG
  * frequent premature ventricular complexes (>1000/24h)
  * non-sustained ventricular arrythmias
  * sustained ventricular arrythmias
  * severe mitral regurgitation
  * myocardial fibrosis with a non-ischemic pattern, especially of papillary muscles and inferolateral wall. The primary endpoint will be considered achieved if at least one of the above mentioned paramentrs will be found in the patient

SECONDARY OUTCOMES:
surgery for mitral valve | 5 years
  occurrence of mitral surgery
sudden cardiac death | 5 years
  occurrence of sudden cardiac death
aborted cardiac arrest | 5 years
  occurrence of aborted cardiac arrest
ventricular arrhythmia | 5 years
  occurrence of non-sustained and/or sustained ventricular tachycardia

CONTACTS AND LOCATIONS:
Overall Officials: Elisabetta Tonet, MD, Principal Investigator — University Hospital of Ferrara
Locations (7):
- Italy (7):
  - University Hospital of Ferrara, Ferrara, Ferrara
  - Cardiology Unit, Bologna
  - Morgagni Hospital, Forlì
  - Cardiology Unit, Palermo
  - Santa Maria delle Croci Hospital, Ravenna
  - Cardiology Unit, Rimini
  - University Hospital fo Trieste, Trieste

IPD SHARING:
Plan to Share IPD: Undecided